CLINICAL TRIAL: NCT00856804
Title: Usefulness of Adding Thalidomide to Peginterferon and Ribavirin in Patients With Hepatitis C and Resistance to Interferon. Phase II
Brief Title: Thalidomide Plus Peginterferon and Ribavirin in Patients With Interferon Resistance
Acronym: TRITAL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Valme University Hospital (Other)
Collaborators: University of Seville (Other)
Responsible Party: Manuel Romero-Gomez, Valme University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRITAL
Record Dates: First submitted 2009-03-03; First posted 2009-03-06 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-03

CONDITIONS: Hepatitis C
Keywords: Thalidomide; Hepatitis C; Interferon resistance; Immunomodulators
MeSH Terms: conditions — Hepatitis C | interventions — Thalidomide; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): thalidomide added to peg-interferon + ribavirina
  Interventions: Drug: thalidomide

INTERVENTIONS:
Drug: thalidomide — Open-label pilot study analyzing the impact of adding thalidomide (200 mg/d)to SOC on 12 weeks virological response in patients with chronic hepatitis C and interferon resistance.
  Other Names: thalidomide adding to peginterferon + ribavirin

SUMMARY:
INDICATION:

Patients with chronic hepatitis C, genotype 1 and non-responders to standard treatment for hepatitis C.

OBJECTIVES:

1. ascertain the rate of sustained response in patients with hepatitis C, genotype 1 with peginterferon + ribavirin resistance.
2. To know the response rate in 12 weeks
3. Describe the tolerance and safety of thalidomide in combination with peginterferon and ribavirin.

DESIGN OF TEST Pilot Study:

The single arm study will:

1. Thalidomide 200 mg and peg-interferon alfa 2b (based on weight: 50-120 mcg / week) + ribavirin (based on weight: 1000-1200mg / day)

Be tracked for 24 weeks after treatment.

Suspended treatment of 12 weeks in patients who have failed a drop of HCV RNA> 2 log.

Patients who have been suspended for any reason, the treatment will be followed during 24 weeks, to assess safety parameters.

SUBJECT NUMBER: 10

ELIGIBILITY:
Inclusion Criteria:

* Men and women in non fertile age.
* HCV RNA detectable in serum.
* Chronic hepatitis C virus with non-cirrhotic compensated liver disease (clinical classification according to Child-Pugh Grade A) (Appendix 1).
* Genotype 1.
* Not responding to treatment with peginterferon alfa-2a in combination with Ribavirin.
* Effective contraceptive measures during treatment and for 6 months after treatment.

Exclusion Criteria:

Patients with any of the following will not be selected for treatment:

* Patients with liver biopsy compatible with cirrhosis F4 Metav classification.
* Patients diagnosed with diabetes or basal glycemia higher than 126 mg / dl
* Women and men of childbearing age
* Treatment with systemic antineoplastic or immunomodulatory (including suprafisiológicas doses of steroids and radiotherapy) 6 months before the first dose of treatment.
* Treatment with any investigational drug 6 weeks before the first dose of treatment.
* History or other evidence of any pathology associated with chronic liver disease than HCV.
* Signs or symptoms of hepatocellular carcinoma.
* History or other evidence of bleeding due to esophageal varices or other conditions consistent with decompensated liver disease.
* neutrophil count <1500 células/mm3 or platelet count <90,000 células/mm3 at Screening.
* Hb <12 g / dL in women or <13 g / dL in men, at the time of evaluation.
* Patients with baseline increased risk of anemia (eg thalassemia, spherocytosis, history of gastrointestinal bleeding, etc.). Or where the presence of anemia would be a medical problem.
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be treated if in the opinion of the investigator, could not tolerate an adequately sharp decline in hemoglobin.
* serum creatinine> 1.5 times above the normal upper limit at the time of valuation.
* History of severe psychiatric illness, particularly depression. Is defined as a serious psychiatric illness requiring treatment with antidepressants or major tranquilizers in therapeutic doses required for major depression or psychosis, respectively, for at least 3 months at any time before or any of the following background: attempted suicide, hospitalization due to of psychiatric illness, or period of disability due to psychiatric illness.
* History of seizure disorder or current use of major anticonvulsants.
* History of immune disease, chronic lung disease associated with limited functionality, serious heart disease, congestive heart failure, advanced atherosclerosis, increased organ transplant or other signs of serious disease, neoplasia, or any other condition deemed by the investigator, prevent the patient is suitable for the study.
* A history of thyroid disease poorly controlled with medications prescribed, elevated concentrations of thyroid stimulating hormone (TSH) with increased thyroid peroxidase antibodies and any clinical manifestation of thyroid disease.
* Pathology involving a risk of acute renal function: dehydration (diarrhea, vomiting), fever, infectious states and / or hypotonic severe (shock, sepsis, urinary infection, neuropathy).
* Evidence of severe retinopathy (eg CMV retinitis, macular degeneration).
* Exploration programanada radiation with intravenous administration of contrast media (IVU, angiography).
* Evidence of drug use in the year prior to study.
* Consumption of alcohol.
* Inability or unwillingness to give informed consent or to comply with the requirements of the study.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Virological response at week 12 | 36 months

SECONDARY OUTCOMES:
Sustained virological response 24 weeks after the end of therapy | 36 months
Safety of using thalidomide together with SOC. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Romero-Gomez, Prof., Principal Investigator — Valme University Hospital
Locations (1):
- Hospital de Valme, Seville, Spain